CLINICAL TRIAL: NCT02646527
Title: Dignity Therapy+: a Brief Psychological and Existential Intervention for Dying Patients and Their Families. A Randomized Controlled Trial
Brief Title: Dignity Therapy+: A Brief Psychological and Existential Intervention for Dying Patients and Their Families.
Acronym: DT-plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss Cancer League (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEK-ZH-2015-0416
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Palliative Care
Keywords: dignity, end of life, existential, treatment
MeSH Terms: conditions — Death | interventions — Dignity Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DT+ (Experimental): Dignity Therapy is conducted with patients and partners
  Interventions: Behavioral: Dignity Therapy
- DT (Experimental): Dignity Therapy is conducted only with patients
  Interventions: Behavioral: Dignity Therapy
- SPC (No Intervention): standard palliative care

INTERVENTIONS:
Behavioral: Dignity Therapy — Dignity Therapy (DT) is a brief psychotherapeutic intervention developed by Chochinov (2012) which has been shown to enhance the end of life experience in people with life-limiting conditions. DT focuses on helping patients with terminal illnesses to go over things that are most meaningful to them and document their legacy. Dignity Therapy+ (DT+) involves patient and partner/family asking questions about their most important achievements, roles and other important aspects of life. DT+ encourages patients saying things to loved ones that have remained unsaid. DT+ consists of 3 sessions (1. introduction (30'); 2. main session (60'), 3. final session (30')) and will be conducted by a trained therapist. All therapy session will be audio-taped, transcribed verbatim by the study coordinator, edited by the therapist and returned to the patient or the patient and partner/family as a 'generativity document'.
  Arms: DT; DT+

SUMMARY:
Background: There has been significant progress in symptom management, pain relief and improvement of quality of life in patients nearing death by implementing palliative care programs. Existential and dignity related issues, such as loss of autonomy and sense of meaning or feeling a burden to others are frequent reasons for psychological distress and desire for hastened death. Dignity Therapy (DT), developed by Chochinov et al., is a brief, individualized psychotherapy for the purpose of relieving distress by directly addressing dignity conserving factors.

Aims: To test whether the inclusion of a patient's partner or designated family member into Dignity Therapy (DT+) could mitigate psychological distress (anxiety and depression) in both, the patient nearing the end of his life experiencing increased psychological distress and the patient's partner/family member compared to the control groups receiving Dignity Therapy in the single setting (DT) or standard palliative care (SPC).

Methods and design: In this randomized controlled trial a total of 159 patients with a diagnosis of an advanced disease and poor prognosis (life expectancy < 6 months) who receive palliative care either in the Palliative Care Centre of the University Hospital Zurich (USZ) or the Clinic Susenberg, Zurich, or in the "Lighthouse" Hospice Zurich, will be randomly assigned to either DT+, DT, or SPC in a 1:1:1 ratio. Patients will be pre-screened and included if they report increased psychological distress (anxiety, depression using the Hospital Anxiety and Depression Scale=HADS). The therapy is guided by trained therapists and consists of 3 audiotaped sessions. The main focus of the intervention is to invite patients to reflect on their most important achievements, roles or other things in their lives or things that they would most want remembered. On completion, the audiorecording is transcribed and edited to provide a clear and readable narrative, the generativity document, which can be passed to a person of the patient's choice. DT+, in contrast to the original intervention developed by Chochinov et al., is a systemic approach in which patient's partners or designated family members are included.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Diagnosis of advanced cancer and life expectancy < 6 months
* Receiving palliative care at the Palliative Care Centre or oncological wards at the University Hospital Zurich, the Susenberg Clinic, or Zurich 'Lighthouse' Hospice
* ≥ 18 years of age
* HADS score ≥ 8

Exclusion Criteria:

* Delirious (ICD-10: F05.9)
* Cognitively impaired
* Too ill to complete the requirements of the protocol
* Unable to speak and read German

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-04; Primary Completion 2021-12 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be psychological distress, as measured by the Hospital Anxiety and Depression Scale (HADS). | 10 days
  questionnaire score

SECONDARY OUTCOMES:
Health related quality of life (HRQol) | 10 days
  questionnaire score

CONTACTS AND LOCATIONS:
Overall Officials: Josef Jenewein, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Devuyst P, Leiter RE, Milliken A, Jenewein J, Blum D, Seiler A. Narrative identity at the end of life: a qualitative analysis of dignity therapy interviews from an existential perspective. BMC Palliat Care. 2025 Oct 23;24(1):269. doi: 10.1186/s12904-025-01876-2. PMID 41131554
- [Derived] Seiler A, Amann M, Hertler C, Christ SM, Schettle M, Kaeppeli BM, Jung-Amstutz J, Nigg C, Pestalozzi BC, Imesch P, Dummer R, Blum D, Jenewein J. Effects of dignity therapy on psychological distress and wellbeing of palliative care patients and family caregivers - a randomized controlled study. BMC Palliat Care. 2024 Mar 14;23(1):73. doi: 10.1186/s12904-024-01408-4. PMID 38486192